CLINICAL TRIAL: NCT03684876
Title: Association Between Renal and Right Cardiac Functions After Urinary Sodium Depletion Following Cardiac Surgery: a Prospective Observational Study
Brief Title: Association Between Renal and Right Cardiac Functions After Urinary Sodium Depletion Following Cardiac Surgery
Acronym: DECONGEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI 2018_843_012
Record Dates: First submitted 2018-07-05; First posted 2018-09-26 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Cardiorenal Syndrome
Keywords: cardiac surgery; venous congestion; diuretic depletion
MeSH Terms: conditions — Cardio-Renal Syndrome; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: diuretic use — use of diuretic

SUMMARY:
Following cardiac surgery, right ventricular function may be altered leading to increase central venous pressure and decrease in renal blood flow. The investigator's standard care includes use of diuretic to avoid interstitial fluid accumulation. The aim of the study is to assess cardiac and renal function before and after depletion by using diuretics

DETAILED DESCRIPTION:
The study will compare cardiac and renal data before and 6 hours after use of diuretic

* Echocardiographic measure of right function (S wave, TAPSE, ventricle surfaces, inferior vena cava diameter) and left function (LVEF, cardiac output
* Renal function: cumulative diuresis, creatinine level variation and incidence of acute kidney injury using KDIGO classification (creatinine level>26.5 or diuresis<0.05 ml kg-1 h-1)

ELIGIBILITY:
Inclusion Criteria:

patient undergoing elective cardiac surgery under cardiopulmonary bypass

Exclusion Criteria:

* heart transplantation
* use of vasopressor
* chronic renal disease (DGF under 30 ml min-1)
* endocarditis
* patient under ECLS or CPIA
* patient under 18-year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient age >=18 years
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
change in renal glomerular filtration before and 6 hours after use of diurectic | at baseline (o hours) and 6 hours after use of diuretic
  change in renal glomerular filtration before and 6 hours after use of diurectic

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No